CLINICAL TRIAL: NCT01077414
Title: Phenomenological Study of Psycho-Socio-Spiritual Healing in the Context of Chronic or Life-Threatening Illness
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 090227; 09-CC-0227
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-11-02

CONDITIONS: Cancer; Pain
Keywords: Psychosocial Functioning; Psychosocial Stress; Palliative Care; Spirituality; Cancer
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* A person s mental state, personal relationships, or spiritual well-being often change in many ways during or after cancer. Some of these changes can have a life-changing positive side, called psycho-socio-spiritual or PSS Healing. For example, a person may feel mentally stronger or more whole than before their cancer.
* Because researchers are interested in enhancing such experiences in other cancer patients, there is interest in developing a way to measure PSS Healing that would be helpful in understanding this phenomenon.

Objective:

- To determine and categorize the characteristics of PSS Healing, which could lead to development of a psychometric instrument to measure it.

Eligibility:

- Adults who have cancer or have had cancer that was diagnosed after the age of 18 and who have had at least one strong positive emotional or mental change in relation to the cancer (e.g., relationships with others, spiritual well-being or faith, thoughts about the meaning of life, reactions to stress).

Design:

* The study design does not involve any treatment or counseling.
* Participants will be interviewed by a research team member. The one-time interview will last up to 2.25 hours and will be audiotaped and transcribed.
* Interviews will consist of an in-depth portion to assess the positive changes in relation to the illness. Participants will then be asked to identify from a list of short descriptions the ones that best reflect their personal experience of PSS Healing.
* Transcribed information will be coded and categorized according to standard research techniques.

DETAILED DESCRIPTION:
We identify healing in the context of chronic or life-threatening illness as a patient-reported outcome consisting of growth or benefit in psychological, social and/or spiritual dimensions representing improvement well above the patient s pre-morbidity baseline. This positive outcome often occurs despite substantial suffering during the illness, even in terminal cases (Kearney 2000).

In previous phenomenological studies, qualitative descriptions of healing and the processes by which it develops have not been structured in categories suitable for the development of a fully validated and standardized psychometric instrument. Also, the relationship of healing to psychometrically measurable constructs such as posttraumatic growth, resilience, coping, and acceptance is not clear.

Objective: This program is to provide (1) a qualitative model of healing-related processes, (2) phenomenological categories of healing suitable for a psychometric instrument development, (3) the relationship of healing to other relevant constructs such as trauma, coping, and adult development, and (4) questionnaire items for healing assessment and (5) software tools that greatly increase the qualitative analysis speed and rigor of phenomenological category building.

Study populations: Two populations of subjects who have experienced a life-threatening disease or serious chronic illness (cancer or cardiac disease) will be recruited from three sites. The first population (50 subjects) are individuals with exemplary healing experiences (life-transforming positive outcomes connected to illness along psychological, social and/or spiritual dimensions) or in the early stages of healing-related processes. In-depth interview data from these subjects will empirically help identify endpoint markers and process pathways of profound healing. The second population (400 subjects) consists of current or past participants in structured healing or medical rehabilitation programs. In a written interview, these participants will qualitatively evaluate questionnaire items for identifying readiness for and progress toward healing using their first-hand, illness-related experience.

Design: This protocol has a qualitative, phenomenological, natural history design similar to identifying features of a medical syndrome or psychological disorder. It has two formats of data collection: in-depth individual interviews of the exemplary healing population, and self-administered written interviews for current participants in formal healing or rehabilitation programs. In-depth interview sessions have 2 1/4-hour duration with three components: a 50-minute, in depth phenomenological interview, a 30-minute short-statement interview (how subjects view healing-related short questionnaire statements), and a 25-minute related-constructs interview (how their positive outcomes, may be related to personality). Interview and short-statement analyses consist of standard qualitative methodologies including transcription, memo-writing, coding, categorization, and modeling.

Outcome measures: None (non-interventional)

ELIGIBILITY:
* INCLUSION CRITERIA FOR ALL SUBGROUPS IN STUDY POPULATION 1:

  1. Physician-diagnosed cancer or cardiac disease.
  2. Audio clarity subjects must be able to participate in oral interviews with sufficient speaking volume and clarity to enable clearly audible recording of the participant s verbal responses using a recorder. For example, subjects with severe hearing disability who nonetheless reads lip well are eligible for enrollment in this study.
  3. Willing to have audio recording during interview subjects must be willing to have the interview recorded with a recorder during oral interviews.
  4. English speaking and reading subjects must be proficient in English speaking and reading. The purpose of the speaking requirement is to aid interview transcription and coding processes. The purpose of the reading requirement is two-fold: (A) for completion of English text documents during enrollment, including written standard psychological exams, with minimal assistance, and (B) fluent reading of specific written text in English is necessary for the training of transcription software to perform automated transcription.
  5. Able to provide informed consent.

SUBGROUP-SPECIFIC INCLUSION CRITERIA IN STUDY POPULATION 1:

1. SFC participants who have completed healing program: have well-established, life-transforming positive psychosocio-spiritual outcome with onset > 6 months before interview
2. SFC-CUP participants who may be considered underserved in healthcare: have well-established, life-transforming positive psychosocio-spiritual outcome with onset > 6 months before interview
3. CRS patients recent cardiac event, beginning rehabilitation: have willingness to participate in a series of face-to-face or telephone interviews
4. CRS patients completed initial 36-session physical rehabilitation: have positive psycho-socio-spiritual outcome with onset after cardiac event
5. NIH CC PPCS patients terminal prognosis or GVHD: positive psycho-socio-spiritual outcome with onset after disease onset or diagnosis

INCLUSION CRITERIA FOR POPULATION 2:

1. Physician-diagnosed cancer.
2. Completion of at least one of the formal programs of palliative care (CC), healing (SFC), or rehabilitation (CRS or CC).
3. No requirement for positive psychological, social, or spiritual change of any duration.
4. English speaking and reading subjects must be proficient in English speaking and reading. The purpose of the speaking requirement is to aid interview transcription and coding processes. The purpose of the reading requirement is two-fold: (A) for completion of English text documents during enrollment, including written standard psychological exams, with minimal assistance, and (B) fluent reading of specific written text in English is necessary for the training of transcription software to perform automated transcription.
5. Able to provide informed consent.

SUBGROUP-SPECIFIC INCLUSION CRITERIA IN STUDY POPULATION 1:

1. SFC participants who have completed healing program: have well-established, life-transforming positive psychosocio-spiritual outcome with onset > 6 months before interview
2. SFC-CUP participants who may be considered underserved in healthcare: have well-established, life-transforming positive psychosocio-spiritual outcome with onset > 6 months before interview
3. CRS patients recent cardiac event, beginning rehabilitation: have willingness to participate in a series of face-to-face or telephone interviews
4. CRS patients completed initial 36-session physical rehabilitation: have positive psycho-socio-spiritual outcome with onset after cardiac event
5. NIH CC PPCS patients terminal prognosis or GVHD: positive psycho-socio-spiritual outcome with onset after disease onset or diagnosis

EXCLUSION CRITERIA FOR THE STUDY POPULATION 1:

1. Age under 18 years. Subjects under 18 years of age are less likely to have a sufficient volume of life experience and maturity of perspective to address the full range and depth of psychological, social and spiritual issues that arise in the context of psycho-socio-spiritual healing.
2. Born with the illness or diagnosed before 17 1/2 years of age. Even if the subject is at least 18 years of age at the time of the interview, the scope of this study is focused on the adult psycho-socio-spiritual response to cancer (see exclusion criterion 1 above).
3. Emotional distress self-report (by the subject) that is equal to or above 3 as indicated on the Distress Thermometer instrument s 0-10 scale.

EXCLUSION CRITERIA FOR POPULATION 2:

1. Age under 18 years. Subjects under 18 years of age are less likely to have a sufficient volume of life experience and maturity of perspective to address the full range and depth of psychological, social and spiritual issues that arise in the context of psycho-socio-spiritual healing.
2. Born with the illness or diagnosed before 17 1/2 years of age. Even if the subject is at least 18 years of age at the time of the interview, the scope of this study is focused on the adult psycho-socio-spiritual response to cancer (see exclusion criterion 1 above).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-09-04; Study Completion 2016-11-02

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Cohen Berger, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Beck CT. The lived experience of postpartum depression: a phenomenological study. Nurs Res. 1992 May-Jun;41(3):166-70. PMID 1584660
- [Background] Beck CT. Teetering on the edge: a substantive theory of postpartum depression. Nurs Res. 1993 Jan-Feb;42(1):42-8. PMID 8424067
- [Background] Beck CT, Gable RK. Postpartum Depression Screening Scale: development and psychometric testing. Nurs Res. 2000 Sep-Oct;49(5):272-82. doi: 10.1097/00006199-200009000-00006. PMID 11009122